CLINICAL TRIAL: NCT04579341
Title: The Effect of Probiotics Supplementation on Glucose Homeostasis, Lipid Profile and Interleukin (IL)-21 and IL-22 Levels in Children With Type 1 Diabetes: A Randomized Placebo-controlled Trial
Brief Title: Probiotics Supplementation Effect on Glucose Homeostasis in Children With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran yousef, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Probiotics
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotics arm (Active Comparator): probiotics administered in addition to insulin regimen
  Interventions: Dietary Supplement: probiotics
- control (No Intervention): regular insulin regimen

INTERVENTIONS:
Dietary Supplement: probiotics — probiotics administration
  Arms: probiotics arm

SUMMARY:
Background: Probiotics influence immune homeostasis, through altering gut microbiota. The efficacy of probiotics in diabetes has been shown in preclinical settings as well as in human trials. Interleukin (IL)-21 and IL22 have been implicated in the pathogenesis of T1D. Objectives: to assess the effect of oral supplementation with probiotics on glycemic control as well as IL-21 and IL-22 levels in children with T1D. Methods: This randomized-controlled trial study included 70 children with T1D. Enrolled children aged 5-18 years with disease duration > 1 year. They were randomly assigned into two groups; intervention group (group A) who received oral probiotics containing Lactobacillus acidophilus La-14 (108 CFU) 0.5 mg once daily. The other group (group B) did not receive any supplementation and served as a control group. Both groups were followed-up for 6 months with assessment of fasting blood glucose (FBG), HbA1c, IL-21 and IL-22 levels.

ELIGIBILITY:
Inclusion Criteria:

* T1D

Exclusion Criteria:

* other types of DM

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2020-10-28 (Estimated); Study Completion 2020-11-10 (Estimated)

PRIMARY OUTCOMES:
glycemic control | 6 months
  HbA1C

CONTACTS AND LOCATIONS:
Overall Officials: Amira Adly, MD, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo, Ramses
  - Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: No